CLINICAL TRIAL: NCT05713396
Title: Long - Term Effect of Quinapril or Losartan or Their Combination on Diabetic Autonomic Neuropathy and Left Ventricular Function Over a Period of 4 Years. A Radionuclide Ventriculography Study.
Brief Title: Diabetic Autonomic Neuropathy and Left Ventricular Function
Acronym: DANEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Matthaios Didagelos, Consultant Cardiologist, AHEPA University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72405
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Quinapril; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quinapril (Q) (Experimental): Patients receiving Quinapril
  Interventions: Drug: Quinapril
- Losartan (L) (Experimental): Patients receiving Losartan
  Interventions: Drug: Losartan
- Quinapril + Losartan (Q+L) (Experimental): Patients receiving both Quinapril and Losartan
  Interventions: Drug: Quinapril + Losartan

INTERVENTIONS:
Drug: Quinapril — Per os
  Arms: Quinapril (Q)
Drug: Losartan — Per os
  Arms: Losartan (L)
Drug: Quinapril + Losartan — Per os
  Arms: Quinapril + Losartan (Q+L)

SUMMARY:
Purpose: To investigate the effect of Quinapril (Q) or Losartan (L) or their combination on definite Diabetic Autonomic Neuropathy (DAN) and left ventricular systolic and diastolic function (LVF) over a period of 4 years.

Patients-methods: Fifty-nine patients with definite DAN [2 or more of the 4 Cardiovascular Reflex Tests (CRTs) were abnormal] were studied for 4 years. Patients were randomly allocated in 3 groups receiving A, 20 mg Q, B, 100 mg L and C, 20 mg Q +100 mg L respectively. CRTs analyzed with Mean Circular Resultant (MCR), Valsalva index, 30:15 ratio and postural hypotension. LV function was investigated with radionuclide ventriculography (RNV) at rest. Ejection fraction was used to assess LV systolic function, while peak filling rate, first third filling fraction, and atrial contribution to ventricular filling were used to investigate LV diastolic function. CRTs and RNV were performed at baseline and after 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Diabetes mellitus
3. Diabetic autonomic neuropathy

Exclusion Criteria:

1. Coronary artery disease
2. Arterial hypertension
3. Heart failure with reduced ejection fraction LVEF<40%
4. Any contraindication to undergo radionuclide ventriculography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
MCR | 4 years
  Mean Circular Resultant
AV | 4 years
  Atrial contribution to ventricular filling

SECONDARY OUTCOMES:
E/I Index | 4 years
  Expiration/Inspiration Index
SD | 4 years
  Standard Deviation
Valsalva Index | 4 years
  Valsalva Maneuver
30:15 Index | 4 years
  Variation of R-R interval during postural change
Postural hypotension | 4 years
  Variation of systolic blood pressure during postural change (standing)
EF | 4 years
  Left ventricular ejection fraction
PER | 4 years
  Peak emptying rate
PFR | 4 years
  Peak filling rate Peak filling rate
1/3 FF | 4 years
  Filling fraction during the first third of the diastole
TPF/FT | 4 years
  Time to peak filling time/filling time

CONTACTS AND LOCATIONS:
Overall Officials: Triantafillos Didangelos, Professor, Principal Investigator — AHEPA University Hospital, Thessaloniki, Greece
Locations (1):
- Diabetes Center, 1st Propeudetic Department of Internal Medicine, Medical School, Aristotle University of Thessaloniki, "AHEPA'' Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No